CLINICAL TRIAL: NCT03808831
Title: Clinical Application of a Fall Detection and Prevention System for Reducing Falls in the Elderly
Brief Title: Fall Detection and Prevention System for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Principal Investigator, I-Hsuan Chen, Assistant professor, Fooyin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGHKS18-CT6-13
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Accidental Falls
Keywords: Fall detection; Fall prevention; Accelerometer; Elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental groups (Experimental): Subjects in the experimental group will wear the fall detection and prevention system on the lower back. The system records near-fall and fall events; meanwhile, it alarms subjects while detecting near-fall events and alarms caregivers while detecting fall events.
  Interventions: Device: Fall detection and prevention system
- Sham group (Sham Comparator): In the sham group, subjects wear a sham system with record but no alert function.
  Interventions: Device: Sham fall detection and prevention system

INTERVENTIONS:
Device: Fall detection and prevention system — The fall detection and prevention system records near-fall and fall events; meanwhile, it alarms subjects while detecting near-fall events and alarms caregivers while detecting fall events.
  Arms: Experimental groups
Device: Sham fall detection and prevention system — The sham system with record but no alert function
  Arms: Sham group

SUMMARY:
There is an urgent need for developing monitoring systems that can detect near-falls and alert persons who suffer from subsequently falls. Therefore, investigators propose a project to study the clinical application of a fall detection and prevention system for reducing falls in the elderly.

The main objectives of the project are to develop the fall detection and prevention system and to investigate its effectiveness in preventing falls for the elderly. Eighty elderly will be recruited and randomly allocated into either the experimental or sham groups (n=40 for each group). Subjects in the experimental group will wear the fall detection and prevention system on the lower back. The system records near-fall and fall events; meanwhile, it alarms subjects while detecting near-fall events and alarms caregivers while detecting fall events. In the sham group, subjects wear a sham system with record but no alert function. Both groups will receive the same treadmill walking training for 30 minutes per session, 3 sessions per week for 6 weeks. The outcome measures including falls, balance function, gait ability, physical activity, and quality of life will be assessed before intervention, after intervention, and at 6-months follow-up.

Fall-induced physiological and psychological consequences limit daily activities and reduce quality of life in the elderly. The proposed study innovates a system that not only detects but also alarms users to prevent falls. Moreover, quantitative measurement of such fall detection and prevention system will be investigated for the elderly in this project. This study provides practical and efficacy solutions to prevent falls for home and community settings.

DETAILED DESCRIPTION:
Fall prevention is the most important issue for the elderly. Due to the low cost and convenience of wearable devices, numerous techniques have been developed to detect falls in clinical environment. However, such effects with large populations have not been established for the elderly. Another, existing systems mainly focus on detecting a fall with little emphasis on fall prediction and prevention. There is an urgent need for developing monitoring systems that can detect near-falls and alert persons who suffer from subsequently falls. Therefore, investigators propose a project to study the clinical application of a fall detection and prevention system for reducing falls in the elderly.

The main objectives of the project are to develop the fall detection and prevention system and to investigate its effectiveness in preventing falls for the elderly. Eighty elderly will be recruited and randomly allocated into either the experimental or sham groups (n=40 for each group). Subjects in the experimental group will wear the fall detection and prevention system on the lower back. The system records near-fall and fall events; meanwhile, it alarms subjects while detecting near-fall events and alarms caregivers while detecting fall events. In the sham group, subjects wear a sham system with record but no alert function. Both groups will receive the same treadmill walking training for 30 minutes per session, 3 sessions per week for 6 weeks. The outcome measures including falls, balance function, gait ability, physical activity, and quality of life will be assessed before intervention, after intervention, and at 6-months follow-up.

Fall-induced physiological and psychological consequences limit daily activities and reduce quality of life in the elderly. The proposed study innovates a system that not only detects but also alarms users to prevent falls. Moreover, quantitative measurement of such fall detection and prevention system will be investigated for the elderly in this project. This study provides practical and efficacy solutions to prevent falls for home and community settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Able to walk independently for at least 5 m with or without the use of stick, quad stick or AFO
* With a history or fear of falls
* Able to follow the commands

Exclusion Criteria:

* With a severe cardiovascular, respiratory, musculoskeletal or neurological disorder

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in numbers of falls | Change from baseline numbers of falls at 6 weeks
  An event which results in a participant coming to rest inadvertently on the ground or floor or other lower level
Changes in numbers of falls | Change from baseline numbers of falls at 6 months
  An event which results in a participant coming to rest inadvertently on the ground or floor or other lower level
Changes in numbers of near-falls | Change from baseline numbers of near-falls at 6 weeks
  A stumble event or loss of balance that would result in a fall if sufficient recovery mechanisms were not activated
Changes in numbers of near-falls | Change from baseline numbers of near-falls at 6 months
  A stumble event or loss of balance that would result in a fall if sufficient recovery mechanisms were not activated
Changes in scores of Fall Efficacy Scale - International | Change from baseline scores at 6 weeks
  Higher scores represent greater the fear of falling (ranging from 16 to 64)

SECONDARY OUTCOMES:
Changes in center of pressures (cm) | Change from baseline postural sway at 6 weeks
  The point where the total sum of a pressure field acts on a body, causing a force to act through that point
Changes in time (second) to perform timed up and go test | Change from baseline time at 6 weeks
  Longer time represents a worse outcome
Changes in scores of Berg Balance Scale | Change from baseline scores at 6 weeks
  Higher values represent a better outcome (ranging from 0 to 56)
Changes of walking speed (cm/s) | Change from baseline speed at 6 weeks
  The speed at which participants choose to walk
Changes in scores of Functional Gait Assessment | Change from baseline scores at 6 weeks
  Higher values represent a better outcome (ranging from 0 to 30)
Changes in scores of Physical Activity Scale for the Elderly | Change from baseline scores at 6 weeks
  Higher scores represent a greater physical activity (ranging from 0 to 793)
Changes is scores of Short-Form-12 Health Survey | Change from baseline scores at 6 weeks
  Score > 50 indicate better physical or mental health than the mean

CONTACTS AND LOCATIONS:
Overall Officials: I-Hsuan Chen, PhD, Principal Investigator — Department of Physical therapy, Fooyin University
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No